CLINICAL TRIAL: NCT06619340
Title: A Case Series Assessing the Clinical Utility of EXPAREL As an Intra-articular Posteromedial Surgeon Administered (IPSA) Block in Patients Undergoing Primary Unilateral Total Knee Arthroplasty
Brief Title: EXPAREL IPSA Block in Knee Arthroplasty
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Campbell Clinic (Other)
Responsible Party: Principal Investigator, William M. Mihalko, Professor, Department of Orthopaedic Surgery and Biomechanical Engineering, Campbell Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-10012-XP
Record Dates: First submitted 2024-07-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pain, Postoperative; Osteo Arthritis Knee
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Group (Experimental): Patients will receive an EXPAREL IPSA block intraoperatively.
  Interventions: Drug: Exparel

INTERVENTIONS:
Drug: Exparel — 20 milliliter (mL) EXPAREL with 20mL bupivacaine hydrochloride (HCL) 0.5% will be expanded. An 18-gauge bevel needle will be introduced through the capsular pocket at 1 to 2cm proximal to the adductor tubercle at the proximal border of the posteromedial femoral condyle. The needle will be angled proximally and posteriorly, and then advanced to contact the posteromedial capsule. A 20mL bolus of the study drug admixture will be administered. The remaining 20mL of the study drug admixture will be administered to the anterior and lateral knee structures with approximately 1 to 1.5mL administered with each stick to the intended area.

SUMMARY:
This is a case series to assess the clinical utility of an Intra-articular Posteromedial Surgeon Administered (IPSA) Block in patients undergoing primary unilateral total knee arthroplasty.

DETAILED DESCRIPTION:
EXPAREL is approved by the Food and Drug Administration (FDA) for use in adults to produce postsurgical regional analgesia via an adductor canal block. The purpose of this study is to evaluate the clinical utility of a surgeon administered EXPAREL adductor canal block intraoperatively in patients undergoing primary unilateral total knee arthroplasty (TKA).

Patients will not be randomized - all patients will receive an EXPAREL IPSA block intraoperatively. Visual Analog Scale, patient reported outcomes, and patient's satisfaction with pain management will be recorded. Adverse events will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Indicated to undergo primary unilateral total knee arthroplasty under spinal anesthesia.
2. Primary indication for TKA is degenerative osteoarthritis of the knee.
3. American Society of Anesthesiologists physical status 1, 2, or 3.
4. Able to provide informed consent, adhere to study schedule, and complete all study assessments.
5. Body Mass Index (BMI) > 18 and < 40 kg/m2.

Exclusion Criteria:

1. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (e.g., amide-type local anesthetics, opioids, bupivacaine HCL, non-steroidal anti-inflammatory drugs (NSAIDs)).
2. Planned concurrent surgical procedure (e.g., bilateral TKA).
3. Undergoing unicompartmental TKA or revision TKA.
4. Concurrent painful physical condition (e.g. arthritis, fibromyalgia, cancer) that may require analgesic treatment with NSAIDs or opioids in the post dosing period for pain that is not strictly related to the knee surgery and which, in the Investigator's opinion, may confound the post dosing assessments.
5. Previous open knee surgery on the knee being considered for TKA. Prior arthroscopy is permitted.
6. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
7. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, could interfere with study assessments or compliance.
8. Currently pregnant, nursing, or planning to become pregnant during the study.
9. Clinically significant medical disease that, in the opinion of the Investigator, would make participation in a clinical study inappropriate. This includes diabetic neuropathy, coagulation or bleeding disorders, severe peripheral vascular disease, renal insufficiency, hepatic dysfunction or other conditions that would constitute a contraindication to participation in the study.
10. Chronic opioid use (average ≥30 oral morphine equivalents/day) within 30 days prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment - 24hr recall | Study Enrollment, Post-operative Day 1, Post-operative Day 2, Post-operative Day 3, Post-operative Day 14, Post-operative Day 42
  On a 0-10 scale, record worst pain in the last 24 hours and average pain in the last 24 hours, with 0 being no pain at all and 10 being the worst pain possible.
Pain Assessment - current pain | Study Enrollment, On Admission to Surgery, on Post Anesthesia Care Unit (PACU) Admission, every 15 minutes from PACU admission to discharge home, 12 hours after surgery, Post-operative Day (POD) 1, POD 2, POD 3, POD 14, POD 42
  On a 0-10 scale, record current pain level, with 0 being no pain at all and 10 being the worst pain possible.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement | Enrollment, Post-operative Day 14, Post-operative Day 42
  Patient reported outcome on overall knee health where 0 represents total knee disability and 100 represents perfect knee health.
Forgotten Joint Score | Post-operative Day 14, Post-operative Day 42
  Patient reported outcome on patient's awareness of their artificial joint. The higher the score, the less aware the patient is about their joint during activities of daily living.
Breakthrough Pain Assessment | In PACU before administration of breakthrough pain medication
  On a 0-10 scale, record current pain score before administration of breakthrough pain medication in PACU where 0 represents no pain at all and 10 represents worst pain possible.
Patient Satisfaction with Pain Management | 12 hours after surgery, Post-operative Day 14, Post-operative Day 42
  On a 0-10 scale, record patient's satisfaction with pain management where 0 represents not satisfied at all and 10 represents very satisfied.

OTHER OUTCOMES:
Temperature | Before study medication administration, upon arrival in PACU, 12 hours after surgery
  Oral temperature will be taken in Fahrenheit
Resting heart rate | Before study medication administration, upon arrival in PACU, 12 hours after surgery
  beats per minute
Blood pressure | Before study medication administration, upon arrival in PACU, 12 hours after surgery
  Systolic and diastolic blood pressure will be measured in millimeter of mercury
Respiratory rate | Before study medication administration, upon arrival in PACU, 12 hours after surgery
  Breath per minute
Oxygen saturation | Before study medication administration, upon arrival in PACU, 12 hours after surgery
  Measured by pulse oximetry in percent
Concomitant medication use | From signing informed consent form through 72 hours post-surgery.
  Any medication use, including opioids and analgesics
Adverse Event | From day of surgery to postoperative day 42
  Any adverse event that patient experiences

CONTACTS AND LOCATIONS:
Overall Officials: William Mihalko, MD, PhD, Principal Investigator — Campbell Clinic
Locations (1):
- Campbell Clinic, Germantown, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No